CLINICAL TRIAL: NCT02858726
Title: A Two-Part, Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Intravenous CR845 in Hemodialysis Patients With Moderate-to-Severe Pruritus
Brief Title: Study to Evaluate IV CR845 in Hemodialysis Patients With Moderate-to-Severe Pruritus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR845-CLIN2101
Record Dates: First submitted 2016-07-29; First posted 2016-08-08 (Estimated); Results first posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Uremic Pruritus
Keywords: Hemodialysis; CR845; Kappa opioid; Anti-itch; difelikefalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CR845 0.5mcg/kg (Experimental): Part A of study: IV CR845 0.5 mcg/kg administered after each dialysis session (3 times/week)
  Interventions: Drug: CR845 0.5 mcg/kg
- CR845 1 mcg/kg (Experimental): Part A of study: IV CR845 1 mcg/kg administered after each dialysis session (3 times/week)
  Interventions: Drug: CR845 1 mcg/kg
- CR845 1.5mcg/kg (Experimental): Part A of study: IV CR845 1.5 mcg/kg administered after each dialysis session (3 times/week)
  Interventions: Drug: CR845 1.5mcg/kg
- Placebo (Placebo Comparator): Part A of study: IV Placebo administered after each dialysis session (3 times/week)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CR845 0.5 mcg/kg — IV medication delivered three times/week
  Other Names: CR845
  Arms: CR845 0.5mcg/kg
Drug: CR845 1 mcg/kg — IV medication delivered three times/week
  Other Names: CR845
  Arms: CR845 1 mcg/kg
Drug: CR845 1.5mcg/kg — IV medication delivered three times/week
  Other Names: CR845
  Arms: CR845 1.5mcg/kg
Drug: Placebo — IV medication delivered three times/week
  Arms: Placebo

SUMMARY:
2 Part Study: Part A will assess 3 different dosing levels of IV CR845 versus placebo in patient on hemodialysis who have moderate-to-severe itching due to uremic pruritus. Patients will receive either CR845 or placebo after each dialysis session for eight weeks. The safety and efficacy of CR845 will be monitored throughout the study. A sub-group of patients will also have pharmacokinetic assessments completed. Part B of the study will assess one dose of IVCR845 versus placebo for 12 weeks in patients on hemodialysis who have moderate-to-severe itching. The dose of CR845 used in Part B will be based on safety and efficacy found in Part A.

DETAILED DESCRIPTION:
This is a two-part study. Patients participating in Part A will be consented and trained on the completion of questionnaires about the severity of itching and overall health. Patients will be required to complete questionnaires during their visits to the dialysis center and also while at home on other days. Results of the screening questionnaires will assess eligibility for the study. Additional laboratory tests and measurements for safety will also be completed during the screening period. Patients meeting all criteria for entry into Part A of the study will be randomized to receive either one of three different doses of CR845 or a placebo. Patients will receive the study drug for eight weeks IV after each hemodialysis treatment (i.e. 3 times per week). Assessments for intensity of itch and safety will also be completed during the 8 week treatment period. When patients have completed treatment, a Follow-up visit will be completed 7 days later.

Patients participating in Part B will be consented and trained on the completion of questionnaires about itching and overall health. Patients will be required to complete questionnaires during their visits to the dialysis center and also while at home on other days. Laboratory tests and measurements for safety will also be completed during the screening period to determine study eligibility. Patients meeting all criteria for entry into Part B of the study will be randomized to receive either CR845 or a placebo. The dose of CR845 used will have been determined based on the safety and efficacy from Part A. Patients will be dosed with either CR845 or placebo for twelve weeks after each hemodialysis treatment (i.e. 3 times per week). Assessments for intensity of itch and safety will be completed during the treatment period also. When patients have completed treatment, a Follow-up visit will be completed 7 days later.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to participating in this study;
2. Able to communicate clearly with the Investigator and staff, able to read, complete questionnaires, and understand the study procedures;
3. Males or females 18 years of age or older;
4. ESRD patients who have been on hemodialysis 3 times per week for at least 3 months prior to the start of Screening;
5. Women of child-bearing potential must have a negative serum pregnancy test and agree to practice an acceptable form of birth control for the duration of the study
6. Male patients that are not biologically or surgically sterile must agree to practice an acceptable from of birth control for the duration of the study
7. Weigh between 88.2 lb (40.0 kg) and 297.6 lb (135.0 kg).
8. Patient must self-report pruritus in the month prior to screening.
9. If patient is receiving treatment for itch, this treatment must be stable prior to screening and during treatment period.
10. At least 2 single-pool Kt/V measurements ≥ 1.2, or at least 2 urea reduction ratio measurements ≥ 65%, or 1 single-pool Kt/V measurement ≥ 1.2 and 1 urea reduction ratio measurement ≥ 65% on different dialysis days during the 3 months period prior to Screening;
11. Patient who self-categorize as moderate-to-severe itch.

Exclusion Criteria:

1. Known to be non-compliant with dialysis treatment (i.e., has missed more than 2 dialysis sessions in the past 2 months because of non-compliance);
2. Anticipated to receive a kidney transplant during the study;
3. Known history of allergic reaction to opiates, such as hives
4. Known or suspected history of alcohol, narcotic, or other drug abuse or dependence within 12 months prior to Screening;
5. Patient has any clinically relevant acute or chronic medical or neuropsychiatric condition which, in the opinion of the Investigator, would pose undue risk to the patient, would impede completion of the study procedures, or would compromise the validity of the study measurements;
6. Serum alanine aminotransferase or aspartate aminotransferase greater than 2.5 times the reference upper limit of normal (ULN), or total bilirubin greater than 2 times ULN at Screening;
7. Received another investigational drug within 30 days prior to the start of Screening or has planned to participate in another clinical trial while enrolled in this study;
8. Has pruritus probably or definitely attributed to a cause other than ESRD or its complications (e.g., patients with concomitant pruritic dermatological disease or cholestatic liver disease would be excluded). (Note: Patients whose pruritus is attributed to ESRD complications such as hyperparathyroidism, hyperphosphatemia, anemia, or the dialysis procedure or prescription may be enrolled);
9. Has localized itch restricted to the palms of the hands;
10. Has pruritus only during the dialysis session (by patient report);
11. Anticipated to receive opioid antagonists (e.g., naloxone, naltrexone), or opioid mixed agonist-antagonist (e.g., buprenorphine, nalbuphine) from the start of Screening through the end of the Treatment Period;
12. Used Salvia divinorum or Salvinorin A within 30 days prior to the start of Screening or is anticipated to use it during the study;
13. Received ultraviolet B treatment within 30 days prior to the start of Screening or anticipated to receive such treatment during the study;
14. Participated in a previous clinical trial with CR845.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2016-06; Primary Completion 2017-03-14 (Actual); Study Completion 2017-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederique Menzaghi, PhD, Study Director — Cara Therapeutics
Locations (26):
- United States (26):
  - Cara Therapeutics Investigator Site, Phoenix, Arizona
  - Cara Therapeutics Study Site, Pine Bluff, Arkansas
  - Cara Therapeutics Investigator Site, Long Beach, California
  - Cara Therapeutics Study Site, Northridge, California
  - Cara Therapeutics Study Site, Whittier, California
  - Cara Therapeutics Study Site, Denver, Colorado
  - Cara Therapeutics Study Site, Hollywood, Florida
  - Cara Therapeutics Study Site, Tampa, Florida
  - Cara Therapeutics Study Site, Winter Park, Florida
  - Cara Therapeutics Study Site, Augusta, Georgia
  - Cara Therapeutics Study Site, Meridian, Idaho
  - Cara Therapetics Study Site, Creve Coeur, Missouri
  - Cara Therapeutics Study Site, Kansas City, Missouri
  - Cara Therapeutics Study Site, Omaha, Nebraska
  - Cara Therapetics Investigator Site, Albuquerque, New Mexico
  - Cara Therapeutics Study Site, Gallup, New Mexico
  - Cara Therapeutics Study Site, College Point, New York
  - Cara Therapeutics Investigator Site, Mineola, New York
  - Cara Therapeutics Investigator Site, Wilmington, North Carolina
  - Cara Therapeutics Study Site, Winston-Salem, North Carolina
  - Cara Therapeutics Study Site, Bethlehem, Pennsylvania
  - Cara Therapeutics Investigator Site, Philadelphia, Pennsylvania
  - Cara Therapeutics Study Site, Chattanooga, Tennessee
  - Cara Therapetics Study Site, Knoxville, Tennessee
  - Cara Therapeutics Study Site, San Antonio, Texas
  - Cara Therapeutics Study Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 226 enrolled participants, 175 met inclusion criteria and were randomized to treatment.
Groups:
- CR845 0.5mcg/kg: IV CR845 0.5 mcg/kg administered after each dialysis session (3 times/week)
- CR845 1 mcg/kg: IV CR845 1 mcg/kg administered after each dialysis session (3 times/week)
- CR845 1.5mcg/kg: IV CR845 1.5 mcg/kg administered after each dialysis session (3 times/week)
- Placebo: IV Placebo administered after each dialysis session (3 times/week)
Period: Overall Study
Arm/Group | CR845 0.5mcg/kg | CR845 1 mcg/kg | CR845 1.5mcg/kg | Placebo
Started | 44 | 42 | 44 | 45
Completed | 39 | 35 | 33 | 42
Not Completed | 5 | 7 | 11 | 3
Not completed — Adverse Event | 4 | 4 | 9 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0
Not completed — Noncompliance | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CR845 0.5mcg/kg | CR845 1 mcg/kg | CR845 1.5mcg/kg | Placebo | Total
Number analyzed (Participants) | 44 | 41 | 44 | 45 | 174
Age, Continuous [Mean (Full Range); unit: years] | 57.9 [29 to 80] | 58.2 [26 to 84] | 54.1 [29 to 74] | 59.0 [27 to 84] | 57.3 [26 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 16 | 17 | 69
  Male | 26 | 23 | 28 | 28 | 105
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2 | 4
  Asian | 2 | 0 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 24 | 22 | 31 | 25 | 102
  White | 17 | 19 | 10 | 16 | 62
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Weekly Mean of the Daily 24-hour Worst Itching Intensity NRS Score During Week 8
Description: Intensity of itch was measured using a numerical rating scale (NRS) used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable". Higher scores meant worse itch intensity.
Time Frame: Baseline, Week 8
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CR845 0.5mcg/kg | CR845 1 mcg/kg | CR845 1.5mcg/kg | Placebo
Number analyzed (Participants) | 44 | 41 | 44 | 45
score on a scale | -3.8 (0.4) | -2.8 (0.4) | -3.2 (0.4) | -1.9 (0.4)
Statistical Analysis 1: Comparison: CR845 0.5mcg/kg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; MMRM with effects for treatment, visit, treatment by visit interaction, and covariates for prior anti-itch medication usage and baseline score; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-2.8 to -0.8], Standard Error of Mean 0.5
Statistical Analysis 2: Comparison: CR845 1 mcg/kg vs Placebo; Test type: Superiority; p = 0.107, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.9 to 0.2], Standard Error of Mean 0.5
Statistical Analysis 3: Comparison: CR845 1.5mcg/kg vs Placebo; Test type: Superiority; p = 0.019, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -1.2, 95% CI 2-sided [-2.3 to -0.2], Standard Error of Mean 0.5

2. Secondary Outcome: Improvement in Itch-related Quality of Life as Assessed by the Change From Baseline in Total Skindex-10 Scale Score at the End of Week 8
Description: The Skindex-10 Scale is a multidimensional questionnaire which assesses itch-related quality of life over the past week. The questions cover 3 domains: disease, mood/emotional distress, and social functioning domain. A lower total score represents better quality of life. The minimum score is 0 and the maximum score is 60 (or total score can range from 0 to 60) with a higher score meaning a worse quality of life.
Time Frame: Baseline, Week 8
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CR845 0.5mcg/kg | CR845 1 mcg/kg | CR845 1.5mcg/kg | Placebo
Number analyzed (Participants) | 44 | 41 | 44 | 45
score on a scale | -18.7 (2.0) | -15.5 (2.2) | -15.1 (2.3) | -8.2 (2.0)
Statistical Analysis 1: Comparison: CR845 0.5mcg/kg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.4, 95% CI 2-sided [-16.0 to -4.8], Standard Error of Mean 2.8
Statistical Analysis 2: Comparison: CR845 1 mcg/kg vs Placebo; Test type: Superiority; p = 0.016, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.2, 95% CI 2-sided [-13.1 to -1.4], Standard Error of Mean 3.0
Statistical Analysis 3: Comparison: CR845 1.5mcg/kg vs Placebo; Test type: Superiority; p = 0.026, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.8, 95% CI 2-sided [-12.8 to -0.8], Standard Error of Mean 3.0

ADVERSE EVENTS:
Time Frame: The period of adverse event reporting started after the signing of the ICF through the study follow-up visit or early termination visit (or 7 days after the last dose if no early termination visit was conducted).
Arm/Group | CR845 0.5mcg/kg | CR845 1 mcg/kg | CR845 1.5mcg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/44 | 0/41 | 2/44 | 1/45
Serious Adverse Events (participants affected / at risk) | 10/44 | 6/41 | 11/44 | 4/45
Other Adverse Events (participants affected / at risk) | 22/44 | 16/41 | 18/44 | 3/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CR845 0.5mcg/kg (N=44) | CR845 1 mcg/kg (N=41) | CR845 1.5mcg/kg (N=44) | Placebo (N=45)
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 2 | 0
Impaired self-care (General disorders) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 3 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Septic embolus (Infections and infestations) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 2
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic ischaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Stenotrophomonas infections (Infections and infestations) | 0 | 0 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CR845 0.5mcg/kg (N=44) | CR845 1 mcg/kg (N=41) | CR845 1.5mcg/kg (N=44) | Placebo (N=45)
Diarrhoea (Gastrointestinal disorders) | 7 | 3 | 4 | 0
Dizziness (Nervous system disorders) | 6 | 3 | 2 | 2
Nausea (Gastrointestinal disorders) | 5 | 1 | 3 | 0
Somnolence (Nervous system disorders) | 2 | 2 | 5 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 2 | 0
Headache (Nervous system disorders) | 0 | 5 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 2 | 3 | 0
Fatigue (General disorders) | 1 | 1 | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 3 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-05-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT02858726/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT02858726/SAP_001.pdf